CLINICAL TRIAL: NCT03472508
Title: A Randomized, Double-Blind, Controlled Trial on the Homocysteine-Lowering Effects of Different Doses of Folic Acid Among Patients With Hypertension According to Methylenetetrahydrofolate Reductase C677T Genotypes
Brief Title: H-Type Hypertension Precision Medicine Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Ausa Pharmed Co.,Ltd (Industry)
Collaborators: Second Affiliated Hospital of Nanchang University (Other); Shenzhen Evergreen Medical Institute (Unknown); Nanfang Hospital, Southern Medical University (Other); Peking University First Hospital (Other); The First People's Hospital of Lianyungang (Other); People's Hospital of Rongcheng (Unknown); Anqing Research Center of Anhui Medical University Biomedical Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ausa1801
Record Dates: First submitted 2018-03-14; First posted 2018-03-21 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Hypertension
Keywords: Folic acid; Homocysteine; MTHFR C677T; RCT; Precision treatment
MeSH Terms: conditions — Hypertension | interventions — Folic Acid; Enalapril

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, double-blind, controlled clinical trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- 0 mg folic acid (Sham Comparator): Enalapril Maleate (10mg) with 0 mg folic acid
  Interventions: Drug: Folic Acid; Drug: Enalapril
- 0.4mg Folic acid (Active Comparator): Enalapril Maleate and Folic Acid Tablets (Yiye) (10mg:0.4mg)
  Interventions: Drug: Folic Acid; Drug: Enalapril Maleate and Folic Acid Tablets (Yiye)
- 0.6mg Folic acid (Active Comparator): Enalapril Maleate and Folic Acid Tablets (Yiye) (10mg:0.4mg) with 0.2 mg folic acid
  Interventions: Drug: Folic Acid; Drug: Enalapril Maleate and Folic Acid Tablets (Yiye)
- 0.8mg Folic acid (Active Comparator): Enalapril Maleate and Folic Acid Tablets (Yiye) (10mg:0.8mg)
  Interventions: Drug: Folic Acid; Drug: Enalapril Maleate and Folic Acid Tablets (Yiye)
- 1.2mg Folic acid (Active Comparator): Enalapril Maleate and Folic Acid Tablets (Yiye) (10mg:0.8mg) with 0.4 mg folic acid
  Interventions: Drug: Folic Acid; Drug: Enalapril Maleate and Folic Acid Tablets (Yiye)
- 1.6mg Folic acid (Active Comparator): Enalapril Maleate and Folic Acid Tablets (Yiye) (10mg:0.8mg) with 0.8 mg folic acid
  Interventions: Drug: Folic Acid; Drug: Enalapril Maleate and Folic Acid Tablets (Yiye)
- 2.0mg Folic acid (Active Comparator): Enalapril Maleate and Folic Acid Tablets (Yiye) (10mg:0.8mg) with 1.2 mg folic acid
  Interventions: Drug: Folic Acid; Drug: Enalapril Maleate and Folic Acid Tablets (Yiye)
- 2.4mg Folic acid (Active Comparator): Enalapril Maleate and Folic Acid Tablets (Yiye) (10mg:0.8mg) with 1.6 mg folic acid
  Interventions: Drug: Folic Acid; Drug: Enalapril Maleate and Folic Acid Tablets (Yiye)

INTERVENTIONS:
Drug: Folic Acid — Folic acid used in this study are listed products. All drugs used in the double-blind treatment period of this study will be loaded into safety capsules with the same outer appearance; all parties involved in the trial will be unaware of the contents of the capsules.
Drug: Enalapril Maleate and Folic Acid Tablets (Yiye) — Enalapril Maleate and Folic Acid Tablets (Yiye) have been approved for listing by the China Food and Drug Administration. Approval number: Zhunzi H20103723.All drugs used in the double-blind treatment period of this study will be loaded into safety capsules with the same outer appearance; all parties involved in the trial will be unaware of the contents of the capsules.
  Arms: 0.4mg Folic acid; 0.6mg Folic acid; 0.8mg Folic acid; 1.2mg Folic acid; 1.6mg Folic acid; 2.0mg Folic acid; 2.4mg Folic acid
Drug: Enalapril — Enalapril used in this study are listed products. All drugs used in the double-blind treatment period of this study will be loaded into safety capsules with the same outer appearance; all parties involved in the trial will be unaware of the contents of the capsules.
  Arms: 0 mg folic acid

SUMMARY:
This is a multicenter, randomized, double-blind, controlled clinical trial. It aims to investigate the effects of different doses of folic acid on lowering homocysteine (Hcy) in patients with hypertension with different genotypes of MTHFR C677T and to determine a dose-response relationship.

This study consists of 3 phases: screening ( 2-10 days ), run-in period (0-2 weeks), and double-blind treatment (8 weeks). Follow-up visits will take place at the beginning of both the run-in period and the double-blind treatment period, and at the end of the 2nd, 4th, 6th, and 8th weeks. Hypertensive patients demonstrating good tolerance and adherence to angiotensin converting enzyme inhibitor (ACEI) drugs and who have already been genotyped for MTHFR C677T polymorphism may pass over the run-in period and directly enter the double-blind randomized treatment period. No medications that could affect the assessment of efficacy may be taken during any stage of the study.

DETAILED DESCRIPTION:
Phase I: Screening（V0）

Phase I takes place for about 2-10 days. The purpose is to obtain informed consent and make a preliminary assessment of the patient.

At the first screening visit (V0), or prior to the official treatment visit, a clinical examination will be performed to determine the patient's clinical diagnosis and to determine eligibility for inclusion in the study. General demographic information and questions related to the inclusion/exclusion criteria of this study will be obtained. Additionally, this will be the time to discuss the impact of participant vacation/travel plans on adherence and compliance with the trial protocol.

Before carrying out any research procedures, the purpose of the study and study procedures will be explained and the participant's informed consent will be obtained.

Clinical Diagnosis and Assessment: Prior to the start of the Run-in Period, baseline data and efficacy evaluation data will be collected according to the study flow chart; blood and urine samples will also be collected.

Blood Pressure Measurement: A unified electronic sphygmomanometer blood pressure measurement will be obtained. Participants will be prohibited from smoking, drinking coffee or tea, and urinating 30 minutes prior. Before taking the measurement, participants will be asked to sit quietly for at least 5 minutes prior; the participant will then be asked to assume a sitting position, with both feet flat on the ground and the upper right arm exposed and at the same height as the heart. After measurement, the sphygmomanometer will display the blood pressure and pulse. The average of 3 consecutive measurements with 1-2 minutes between each measurement will be taken and recorded. The median of 3 pulse measurements will also be recorded.

Laboratory Tests: Female participants of childbearing age must undergo a pregnancy test prior to the run-in period. Based on clinical indications, the investigator may also decide to conduct a pregnancy test at any time throughout the trial as needed. All participants will be asked to complete the following laboratory tests: 12-lead ECG, urinalysis, blood biochemistry, folate, and Hcy assessment during the screening period. All results will be obtained prior to the run-in period visit.

Phase Ⅱ: Run-in Period (V1-V2)

All eligible patients will begin a treatment of enalapril (10mg/d) for a 0 to 2-week open induction period, during which time other antihypertensive drugs may also be concurrently used. MTHFR C677T genotype will also be determined during this phase. The primary purpose of this phase is to assess participant compliance to the enalapril treatment regimen as well as to observe the participant's tolerance to enalapril, so as to avoid including those participants with poor compliance or intolerance to enalapril to the double-blind treatment phase.

Newly diagnosed hypertensives should be given enalapril during the run-in period and can be given other antihypertensive drugs at the clinician's discretion. For hypertensive patients currently using medication, if not currently using enalapril, the clinician should, based on the patient's medical condition, add or switch the patient's medication to enalapril.

Hypertensive patients demonstrating good tolerance and adherence to angiotensin converting enzyme inhibitor (ACEI) drugs and who have already been genotyped for MTHFR C677T polymorphism may pass over the run-in period and directly enter the double-blind randomized treatment period.

Phase Ⅲ: Double-Blind Treatment (V2-V6)

The third phase consists of 8 weeks of a randomized, double-blind treatment. Patients who remain eligible for participation in the study will first be stratified by gender and MTHFR C677T genotype (CC, CT, TT), for a total of 6 strata at the start of V2. Each of the 6 strata will then be randomized into 8 treatment groups: either enalapril only (10mg), or one of the other 7 treatment combinations with various doses of folic acid. During the 8-week double-blind treatment period, other antihypertensive drugs can be combined with the treatment drug to achieve blood pressure control; the patient will be followed-up every 2 weeks during the treatment period, and the treatment drug will be distributed at each visit. During this period, participants should continue to avoid taking medications that may interfere with the evaluation of treatment efficacy.

For participants who complete the run-in period and are eligible to remain in the study, a randomized treatment allocation list will be generated using a stratified, block-wise, randomized approach by MTHFR C677T genotype and gender. This list will assign a unique study ID to every study participant. The ID corresponds to a specific treatment allocation; this ID assignment determines the treatment type the participant will receive.

This study will use a two-level blinding procedure. The first level of blinding will generate a randomized sequence table corresponding each study ID to one of the eight different treatment groups. Each treatment will be given a treatment group code (from a to h) so that the actual treatment cannot be identified from this table. The second level of blinding will denote the type of treatment that corresponds to each of the eight different coded treatment groups (a through h) that were generated from the first level of blinding. The randomized ID's will be generated by a statistical analysis group; the blinding program and all electronic documents regarding the level one and two blinding will be sealed in separate envelopes and protected by the sponsor. The seal cannot be broken before the trial officially undergoes the unblinding process. In addition, the research drug management center will maintain a copy of the treatment allocation list and will be responsible for encoding the treatment drugs and dispensing the medications to the participants based on the treatment allocation list.

ELIGIBILITY:
Inclusion Criteria for run-in period:

* （1）≥ 45 years old;
* （2）A diagnosis or previous diagnosis of essential hypertension, including anyone currently taking antihypertensive drugs; or for those who have not taken antihypertensive drugs within the last 2 weeks, two consecutive examinations were conducted at least one day apart, and both sitting blood pressure (mean value of 3 measurements) met the following criteria: diastolic blood pressure (DBP) ≥90 mmHg or systolic blood pressure (SBP) ≥140 mmHg (the second blood pressure was measured at V1);
* （3）If a study participant is a woman of childbearing age, she agrees to use a reliable contraceptive method during the trial;
* （4）Voluntarily participates and has signed an informed consent form.

Inclusion Criteria for Double-Blind Treatment Period:

* （1）Completed MTHFR C677T gene polymorphism detection in run-in period or MTHFR C677T genotype already known in advance;
* （2）Exhibited good tolerance to enalapril and good overall medication compliance (>80%) in run-in period or previously exhibited good tolerance and adherence to ACEI drugs in previous medication history.
* （3）Voluntarily continues to participate in this study.

Exclusion Criteria:

Participants meeting any of the following criteria may not participate in this study:

* （1）Women who are pregnant and/or lactating; or women who intend to conceive within a year;
* （2）History of allergies to enalapril, folic acid or other components of the compound drug;
* （3）History of adverse reactions or intolerance to enalapril or other ACE inhibitors, or drugs or supplements containing folic acid;
* （4）Diagnosis or suspicion of secondary hypertension;
* （5）Known serious medical conditions, including: Cardiovascular: patients with clinically diagnosed cardiac dysfunction (NYHA class III and above), hypertrophic obstructive cardiomyopathy, clinically significant valvular heart disease, acute coronary syndrome within the last 3 months, or percutaneous coronary intervention (PCI), or coronary artery bypass graft (CABG); or abnormal pre-enrollment ECG test results with clinically significant arrhythmias (atrial flutter, atrial fibrillation, grade II-III atrioventricular block, etc.); Digestive: a previous diagnosis of various types of viral hepatitis that are still in the active phase; abnormal pre-enrollment liver function test results (ALT, AST, GGT, TBIL, or DBIL 3 times higher than normal, ALB ≤ 30g/L); gastrectomy and/or gastrojejunostomy; gastrointestinal dysfunction; Urinary: pre-enrollment serum creatinine greater than 200μmol/L; clinical diagnosis of renal artery stenosis, isolated kidney, kidney transplantation and/or other diseases; Endocrine: type 1 diabetes or uncontrolled type 2 diabetes (fasting blood glucose above 11.1 mmol/L at pre-enrollment); previous diagnosis of hyperthyroidism and failure to correct; Respiratory: pulmonary heart disease; chronic obstructive pulmonary disease; Neuropsychiatric: recent transient ischemic attack or stroke (within the last 3 months); peripheral or severe autonomic dysfunction; mental or nervous system dysfunction, inability to express desire; known drug or alcohol dependence; Malignancy, malnutrition, hematopoietic disorders and other serious diseases.
* （6）Significant signs of abnormalities as seen in laboratory tests or physical characteristics, which, at the discretion of the investigators, indicates that the patient is experiencing a serious illness or, may affect the observation and evaluation of the drug's efficacy or adverse events, or renders the patient unsuitable for participating in this study;
* （7）Patients currently taking folate, B12, or B6, or any compounds containing them, who express an inability or a refusal to stop usage;
* （8）Regular usage of folic acid supplements or compounds containing folic acid in the past 3 months;
* （9）Participation in a clinical trial for a drug that has not yet been officially approved for marketing within one month prior to the first visit.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 3600 (Estimated)
Dates: Start 2018-03-20 (Actual); Primary Completion 2019-03-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage decrease in blood homocysteine levels by the end of the 8th week from baseline. | by the end of the 8th week from the baseline
  Hcy percent decrease =（baseline Hcy - end Hcy) /baseline Hcy *100%

SECONDARY OUTCOMES:
Magnitude of decrease in blood homocysteine by the end of the 8th week from baseline. | by the end of the 8th week from the baseline
  Absolute Hcy reduction (μmol/L) = baseline Hcy - end Hcy
Percentage of increase in blood folate levels by the end of the 8th week from baseline. | by the end of the 8th week from the baseline
  Folate increase rate=(end folate- baseline folate)/baseline folate *100%
  folate increase magnitude= end folate - baseline folate
Magnitude of increase in blood folate levels by the end of the 8th week from baseline. | by the end of the 8th week from the baseline
  Absolute folate reduction (μmol/L)= baseline folate - end folate

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoshu Cheng, MD, Principal Investigator — Second Affiliated Hospital of Nanchang University
Locations (5):
- China (5):
  - Anqing Research Center of Anhui Medical University Biomedical Institute, Anqing, Anhui
  - Peking University First Hosptial, Beijing
  - The First People's Hospital of Lianyungang, Lianyungang
  - Second Affiliated Hospital of Nanchang University, Nanchang
  - People's Hospital of Rongcheng, Rongcheng

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kjeldsen SE, Julius S, Hedner T, Hansson L. Stroke is more common than myocardial infarction in hypertension: analysis based on 11 major randomized intervention trials. Blood Press. 2001;10(4):190-2. doi: 10.1080/08037050152669684. No abstract available. PMID 11800055
- [Background] Collaboration HLT. Lowering blood homocysteine with folic acid based supplements: meta-analysis of randomised trials. Homocysteine Lowering Trialists' Collaboration. BMJ. 1998 Mar 21;316(7135):894-8. PMID 9569395
- [Background] Homocysteine Lowering Trialists' Collaboration. Dose-dependent effects of folic acid on blood concentrations of homocysteine: a meta-analysis of the randomized trials. Am J Clin Nutr. 2005 Oct;82(4):806-12. doi: 10.1093/ajcn/82.4.806. PMID 16210710
- [Background] Wilcken B, Bamforth F, Li Z, Zhu H, Ritvanen A, Renlund M, Stoll C, Alembik Y, Dott B, Czeizel AE, Gelman-Kohan Z, Scarano G, Bianca S, Ettore G, Tenconi R, Bellato S, Scala I, Mutchinick OM, Lopez MA, de Walle H, Hofstra R, Joutchenko L, Kavteladze L, Bermejo E, Martinez-Frias ML, Gallagher M, Erickson JD, Vollset SE, Mastroiacovo P, Andria G, Botto LD. Geographical and ethnic variation of the 677C>T allele of 5,10 methylenetetrahydrofolate reductase (MTHFR): findings from over 7000 newborns from 16 areas world wide. J Med Genet. 2003 Aug;40(8):619-25. doi: 10.1136/jmg.40.8.619. No abstract available. PMID 12920077
- [Background] Xu X, Li J, Sheng W, Liu L. Meta-analysis of genetic studies from journals published in China of ischemic stroke in the Han Chinese population. Cerebrovasc Dis. 2008;26(1):48-62. doi: 10.1159/000135653. Epub 2008 May 30. PMID 18511872
- [Background] Dong Q, Tang G, He M, Cai Y, Cai Y, Xing H, Sun L, Li J, Zhang Y, Fan F, Wang B, Sun N, Liu L, Xu X, Hou F, Shen H, Xu X, Huo Y. Methylenetetrahydrofolate reductase C677T polymorphism is associated with estimated glomerular filtration rate in hypertensive Chinese males. BMC Med Genet. 2012 Aug 16;13:74. doi: 10.1186/1471-2350-13-74. PMID 22897803
- [Background] Huang X, Li Y, Li P, Li J, Bao H, Zhang Y, Wang B, Sun N, Wang J, He M, Yin D, Tang G, Chen Y, Cui Y, Huang Y, Hou FF, Qin X, Huo Y, Cheng X. Association between percent decline in serum total homocysteine and risk of first stroke. Neurology. 2017 Nov 14;89(20):2101-2107. doi: 10.1212/WNL.0000000000004648. Epub 2017 Oct 13. PMID 29030456
- [Result] Qin X, Li J, Cui Y, Liu Z, Zhao Z, Ge J, Guan D, Hu J, Wang Y, Zhang F, Xu X, Wang X, Xu X, Huo Y. MTHFR C677T and MTR A2756G polymorphisms and the homocysteine lowering efficacy of different doses of folic acid in hypertensive Chinese adults. Nutr J. 2012 Jan 10;11:2. doi: 10.1186/1475-2891-11-2. PMID 22230384
- [Result] Qin X, Li J, Cui Y, Liu Z, Zhao Z, Ge J, Guan D, Hu J, Wang Y, Zhang F, Xu X, Wang X, Xu X, Huo Y. Effect of folic acid intervention on the change of serum folate level in hypertensive Chinese adults: do methylenetetrahydrofolate reductase and methionine synthase gene polymorphisms affect therapeutic responses? Pharmacogenet Genomics. 2012 Jun;22(6):421-8. doi: 10.1097/FPC.0b013e32834ac5e8. PMID 21869730
- [Result] Qin X, Li J, Zhang Y, Ma W, Fan F, Wang B, Xing H, Tang G, Wang X, Xu X, Xu X, Huo Y. Prevalence and associated factors of diabetes and impaired fasting glucose in Chinese hypertensive adults aged 45 to 75 years. PLoS One. 2012;7(8):e42538. doi: 10.1371/journal.pone.0042538. Epub 2012 Aug 3. PMID 22880024
- [Result] Huo Y, Li J, Qin X, Huang Y, Wang X, Gottesman RF, Tang G, Wang B, Chen D, He M, Fu J, Cai Y, Shi X, Zhang Y, Cui Y, Sun N, Li X, Cheng X, Wang J, Yang X, Yang T, Xiao C, Zhao G, Dong Q, Zhu D, Wang X, Ge J, Zhao L, Hu D, Liu L, Hou FF; CSPPT Investigators. Efficacy of folic acid therapy in primary prevention of stroke among adults with hypertension in China: the CSPPT randomized clinical trial. JAMA. 2015 Apr 7;313(13):1325-35. doi: 10.1001/jama.2015.2274. PMID 25771069
- [Derived] Huang X, Bao H, Ding C, Li J, Cao T, Liu L, Wei Y, Zhou Z, Zhang N, Song Y, Chen P, Jiang C, Xie L, Qin X, Zhang Y, Li J, Sun N, Tang G, Wang X, Wang H, Huo Y, Cheng X; Precision Folic Acid Trial to lower homocysteine (PFAT-Hcy) Trial Investigators. Optimal folic acid dosage in lowering homocysteine: Precision Folic Acid Trial to lower homocysteine (PFAT-Hcy). Eur J Nutr. 2024 Aug;63(5):1513-1528. doi: 10.1007/s00394-024-03344-8. Epub 2024 Mar 13. PMID 38478042
- [Derived] Chen P, Tang L, Song Y, Wang B, Qin X, Zhang N, Wei Y, Xu X, Zhou Z, He Q, Liu L, Siddiqi SM, Huang X, Cheng X, Tang G, Duan Y, Zhou H, Jiang J, Li S. Association of folic acid dosage with circulating unmetabolized folic acid in Chinese adults with H-type hypertension: a multicenter, double-blind, randomized controlled trial. Front Nutr. 2023 Sep 14;10:1191610. doi: 10.3389/fnut.2023.1191610. eCollection 2023. PMID 37781132